CLINICAL TRIAL: NCT03113864
Title: Beneficial Effects of Lutein on Visual Function in Healthy Subjects
Brief Title: Effects of Lutein on Visual Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting Issue
Sponsor: Kemin Foods LC (Industry)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16-004
Record Dates: First submitted 2017-03-15; First posted 2017-04-14 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2017-04

CONDITIONS: Healthy; Nutrition Poor
Keywords: Vision; Eye Health; Lutein; Carotenoids
MeSH Terms: conditions — Malnutrition | interventions — Lutein

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Parallel Intervention Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties involved in the study are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Will be identical looking to treatment
  Interventions: Dietary Supplement: Placebo
- Lutein (Experimental): 10 mg of FloraGLO Lutein
  Interventions: Dietary Supplement: Lutein

INTERVENTIONS:
Dietary Supplement: Placebo — Daily supplementation for 9 months
  Arms: Placebo
Dietary Supplement: Lutein — Daily Supplementation for 9 months
  Arms: Lutein

SUMMARY:
Randomized, double blind, placebo-controlled intervention trial on the ocular benefits and inflammatory markers improvements of taking FloraGLO Lutein for 9 months. The population of interest is middle-aged men and women who have low levels of carotenoids in their eyes.

DETAILED DESCRIPTION:
The participants will be given a brief explanation of the study and asked to sign an informed consent form. During the screening visit, pre-study parameters will be measured in order to assess the subjects' eligibility to participate.

These include:

1. Medical History
2. Vital signs, Height and weight and BMI calculation
3. Visual Parameters
4. Blood draw for clinical chemistry and hematological safety

Intervention Period:

At baseline visual parameters and a serum sample for analysis of inflammatory markers will be taken. Supplements will be dispensed. Study visits will then be conducted every 3 months. At these visits, subjects will have visual parameters, adverse events, study diary, vitals, a questionnaire evaluating health/diet/exercise/alcohol, product distribution and compliance checked. A final serum/plasma sample will be taken at the final visit for re-assessment of safety parameters and inflammatory markers.

Compliance check:

The number of tablets dispensed at baseline and returned, as well as all intake information from a subject diary. Per protocol population is defined apriori as >80%.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 40-60 years
* Corrected Visual Acuity of 20/20 to 20/25
* MPOD 0.05- 0.30 OD units
* Must be able to give written informed consent in English
* BMI < or = 30 kg/m2
* Subject is willing to maintain a habitual diet and physical activity patterns throughout the study period

Exclusion Criteria:

* Use of carotenoid, fish oil, or n-3 fatty acid supplements (within 2 months of study start)
* Ocular pathologies
* History of active small bowel disease or resection
* Uncontrolled hypertension
* Diabetes mellitus
* Pancreatic disease
* Pregnancy (or planning to become pregnant) or lactation
* Diseases that interfere with fat absorption
* Medication or supplements that contain a significant level of carotenoids
* Medications that interfere with fat absorption
* Use of drugs suspected of interfering with metabolism of blood clotting
* Chronic alcohol intake
* Stroke, head injury with loss of consciousness or seizures
* Severe Amblyopia resulting in visual acuity worse than 0.4 MAR
* Subject is a heavy smoker (> 1 pack/day)
* A regular consumer of lutein rich foods or lutein supplements
* A regular consumer of foods high in DHA intake or DHA supplements
* Subject has donated more than 300 mL of blood during the last three months prior to screening

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Co-primary outcome: Cone Sensitivity Recovery | 9 months
  Visual Parameter
Co-primary outcome: Chromatic Contrast Sensitivity | 9 months
  Visual Parameter

SECONDARY OUTCOMES:
Dark Adaption | 9 months
  Visual Parameter
Macular Pigment Optical Density | 9 months
  Visual Parameter
Visual Acuity | 9 months
  Visual Parameter
Complement Factor D, C5a, and MAC | 9 months
  Inflammatory Marker
Plasma Carotenoid Levels | 9 months
  Blood Marker

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Manchester, Manchester, United Kindgom, United Kingdom

IPD SHARING:
Plan to Share IPD: No